CLINICAL TRIAL: NCT04344574
Title: Serum Level of IL31,33 and 36 in Egyptian Paients With Psoriasis in Assiut University Hospital : Case Control Study
Brief Title: Serum Level of IL31,33 and 36 in Egyptian Paients With Psoriasis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Fatma Elzahraa Adel Ismail, Principal Investigator, Assiut University
Other Study IDs: interleukins in psoriasis
Record Dates: First submitted 2020-04-01; First posted 2020-04-14 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Psoriasis
Keywords: interleukine 31,33 and 36
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Evaluating Serum Level Of IL 31 , IL33 and IL36 and Their Correlation with Disease Activity In Patients With Psoriasis In Assuit University Hospital .

* To correlate their levels with disease activity using PASI score .
* To allow better understanding of the pathophysiological mechanism of the disease .

DETAILED DESCRIPTION:
Serum samples will be collected from 45 psoriasis patients and 45 matched healthy individuals. After full history taking and dermatological examination, the disease severity will be assessed using the psoriasis area and severity index (PASI) score. All patients enrolled in our study had no other autoimmune or systemic diseases and underwent no systemic treatment including glucocorticoids, immunosuppressive drugs, or phototherapy at least 1 month before the PASI score evaluation and sample collection period. Wriiten informed consent will be obtained from all the patients and healthy controls.

Assessment of serum interleukin-31 ,33 and 36 concentrations in psoriatic patients Patients and controls Blood samples will collected from psoriatic patients and controls, and will centrifuged for 15 min at 1000 rpm. Next, the serum samples will be subdivided into small aliquots to be stored at -80°C until analysis for cytokine levels. ELISA kits will be used to determine serum IL-31 , 33 and 36

ELIGIBILITY:
Inclusion Criteria:

* Patients with all types of psoriasis.
* healthy volunteers without a family history of psoriasis or other autoimmune disease.

Exclusion Criteria:

* other autoimmune , other chronic inflammatory or systemic diseases.
* cases received glucocorticoids, immunosuppressive drugs at least 1 month before sample collection .

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: study will be performed on 45 psoriasis patients and 45 healthy matched volunteers without a family history of psoriasis and other autoimmune as well as inflammatory diseases and underwent no systemic treatment including glucocorticoids, immunosuppressive drugs, or phototherapy at least 1 month before the PASI score ,evaluation and sample collection period . All patients will be recruited from the Psoriasis Clinic in Dermatology Department of Assuit University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
describe the serum levels of IL31, IL33 and IL36 in egyptian patients with psoriasis. | Baseline
  1. Blood samples will collected from psoriatic patients and controls.
  2. using ELISA kits to measure serum concentration of IL31 [pg/ml] , IL33 [pg/ml] and IL36 [pg/ml] .
  3. p value less than 0,05 reflect significant increase in serum levels of measured interleukins.
4. Knowing the extent of disease activity by Psoriasis Area and Severity Index (PASI) score. | Baseline
  assessment of the severity of lesions and the area affected into a single score in the range 0 (no disease) to 72 (maximal disease).

SECONDARY OUTCOMES:
serum level of interleukins reflect severity of disease and represent anovel target for antipsoriatic drug theraby. | Baseline
  increase of the serum level of interleukins during disease activity means significant increase which has a value in drug therapy of psoriasis . and vice versa.